CLINICAL TRIAL: NCT00849589
Title: Computerized Screening and Brief Physician Advice to Reduce Teen Drinking
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant application was not funded
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cambridge Health Alliance (Other); Dartmouth-Hitchcock Medical Center (Other); Fallon Clinic (Industry); Tufts Medical Center (Other); University of Vermont (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PA-07-406
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Abuse; Risk Behavior
Keywords: Screening; Brief intervention; Underage drinking
MeSH Terms: conditions — Alcoholism; Risk-Taking; Underage Drinking | interventions — Mass Screening; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Treatment as Usual (TAU)
- 2 (Experimental): Computerized Screening and Brief Physician Advice (SBA)
  Interventions: Behavioral: Computerized screening and brief physician advice
- 3 (Experimental): Computerized screening and brief physician advice with technological extenders (SBA/TE)
  Interventions: Behavioral: Computerized SBA with technological extenders

INTERVENTIONS:
Behavioral: Computerized screening and brief physician advice — Participants complete screening for alcohol use and other health risk behaviors on the computer, receive some related health information on the computer, and meet with a primary care provider for a short discussion of health risk behaviors
  Other Names: Screening; Brief advice; Brief intervention; Underage drinking
  Arms: 2
Behavioral: Computerized SBA with technological extenders — Participants complete screening for alcohol use and other health risk behaviors on the computer, receive some related health information on the computer, and meet with a primary care provider for a short discussion of health risk behaviors. In addition, the provider sends them a brief email or text message at 4 months and 9 months after study entry to reinforce the brief advice.
  Other Names: Screening; Brief advice; Brief intervention; Underage drinking
  Arms: 3

SUMMARY:
The goal of this project is to adapt a computerized Screening and Brief Advice (SBA) protocol that has demonstrated efficacy in reducing underage drinking among adolescent primary care patients and then to test it in a multi-site randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The specific aims of the proposed multisite RCT are:

1. To establish the efficacy of the computerized SBA protocol on alcohol use, on DWI/RWID, and other alcohol-related health risk behaviors;
2. To test the effect of Technological Extenders (TE) on prolonging the beneficial effects of the SBA protocol;
3. To identify moderators, mediators, and optimal responders to the SBA/TE interventions;
4. To examine the association between cessation of underage drinking and other health-risk behaviors in an adolescent primary care sample.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 years old
* patients arriving for routine medical care
* provide informed assent (for those <18) or informed consent (for those 18-21)

Exclusion Criteria:

* medically or psychologically unstable at time of visit
* receiving behavioral health services
* cannot read or understand English at a 6th grade reading level
* unavailable for follow-up assessments

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Initiation of underage drinking | Baseline, 3-months, 6-months, 12-months

SECONDARY OUTCOMES:
Cessation of underage drinking | Baseline, 3-months, 6-months, 12-months

CONTACTS AND LOCATIONS:
Overall Officials: John R. Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Adolescent Substance Abuse Research — http://www.ceasar.org